CLINICAL TRIAL: NCT05129618
Title: A Randomized, Double Blind, Placebo Controlled Tolerability Study of Panosyl Isomaltooligosaccharides (PIMO), in Subjects With Chronic Idiopathic Constipation (CIC)
Brief Title: Tolerability Study of Panosyl Isomaltooligosaccharides (PIMO), in Subjects With Chronic Idiopathic Constipation (CIC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microbiome Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MHS-1031-01
Record Dates: First submitted 2021-10-01; First posted 2021-11-22 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Constipation Chronic Idiopathic
Keywords: CIC; microbiome; PIMO; Panosyl-isomaltooligosaccharides; prebiotic

STUDY DESIGN:
Intervention Model Description: Approximately 200 subjects with CIC who meet all eligibility criteria will be randomized in a 1:1 ratio, with equal numbers of each in each successive group of 50 subjects, to receive either MHS 1031 [1 g (1.4 ml) per day] or 1.4 ml of placebo (1:1) for 8 weeks (Product/Placebo Phase). Upon completion of the 8 week Product/Placebo Phase, Subjects will enter a 4 week open label Product Phase, during which all subjects will receive MHS 1031.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Product Tolerability Arm (Active Comparator): active product: MHS 1031 Panosyl-isomaltooligosaccharides liquid 1 g (1.4 ml) per day
  Interventions: Dietary Supplement: MHS 1031
- Placebo Tolerability Arm (Placebo Comparator): Placebo liquid 1 g (1.4 ml) per day
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: MHS 1031 — prebiotic syrup in individual sachets containing 1g (1.4 ml) of panosyl-isomaltooligosaccharides
  Arms: Product Tolerability Arm
Other: placebo — liquid combination formulation of Neotame 7.92 mcg/g, phosphoric acid, and sterile water, designed to have the same degree of sweetness as the test material, provided in individual sachets containing 1.4 ml.
  Arms: Placebo Tolerability Arm

SUMMARY:
This is a randomized, double blind, placebo controlled trial to evaluate the tolerability of MHS 1031. Tolerability will be assessed using the change in complete spontaneous bowel movements (CSBM), PRO questionnaires, concomitant medication assessments, and assessment of adverse events, from baseline (determined during Screening Phase) to Week 8 (Day 56). The primary analysis will be conducted to assess the tolerability of MHS 1031 product and of the formulated placebo in randomized subjects with CIC diagnosed according to a modified Rome IV criteria.

DETAILED DESCRIPTION:
This study will be conducted as a multicenter, randomized, double blind, placebo controlled trial to evaluate the tolerability of MHS 1031 and tolerability of the formulated placebo. The study consists of a screening phase to establish eligibility and baseline values, followed by 3 distinct study periods.

Subjects with CIC will be determined eligible for the study based on modified Rome IV criteria during a 2 week Screening Phase. Approximately 200 subjects with CIC who meet all eligibility criteria will be randomized in a 1:1 ratio, with equal numbers of each in each successive group of 50 subjects, to receive either MHS 1031 [1 g (1.4 ml) per day] or 1.4 ml of placebo (1:1) for 8 weeks (Product/Placebo Phase). Upon completion of the 8 week Product/Placebo Phase, Subjects will enter a 4 week open label Product Phase, during which all subjects will receive MHS 1031. Subjects who complete the study will enter a 2-week Follow-up Phase, during which subjects will take neither placebo nor MHS 1031.

During the study, tolerability will be assessed on the basis of Patient Reported Outcomes (PRO questionnaires), concomitant medication assessments, and assessment of adverse events. Tolerability is defined as no overall worsening of constipation measurement scores after 8 weeks of taking the product or the placebo compared to baseline scores.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to participate in the study for the required duration, understand and provide signed informed consent, and agrees to undergo all protocol activities.
2. Subject is proficient in reading, writing, and speaking English.
3. Subject is able to complete all required electronic Daily Bowel Movement and Symptoms Questionnaire, daily medication reconciliation surveys (Screening, Product Phase, and Product/Placebo Phase), bi-weekly PAC-SYM and PAC QOL questionnaire, and monthly Study Participant Global Assessment questionnaire entries during the 2 week Screening Phase assessment period and for the duration of the study (ie, the 8 week randomized Product/Placebo Phase, 4 week open label Product Phase and the 2 week Follow up Phase).
4. Males or females between 18 and 75 years of age (inclusive), with a BMI ≥ 19 and < 35 kg/m2. Females must not be pregnant or lactating.
5. Female Subjects of non childbearing potential whether surgically sterile or postmenopausal.
6. Females who are still menstruating must be able to differentiate the abdominal symptoms associated with CIC from those associated with their menses (otherwise protocol assessments of these symptoms may be confounded).
7. Male and female Subjects of childbearing potential must agree to use adequate contraception from the time of informed consent to 2 weeks after receiving the last dose of study product.
8. Subject meets the Rome IV functional constipation criteria as modified for this study for ≥ 3 months prior to the Screening Call. The Rome IV criteria as modified for this study, requires the following:

   1. Subject reports that loose stool is rarely present without the use of laxatives.
   2. Subject does not meet the Rome IV criteria for IBS C.
   3. Subject does not use manual maneuvers (eg, digital evacuation, support of the pelvic floor) to facilitate defecations.
   4. Subject reports a history of < 3 complete spontaneous bowel movements per week.
   5. Subject reports ≥ 2 of the following:

   i. Straining during ≥ 25% of defecations ii. Lumpy or hard stool in ≥ 25% of defecations iii. Sensation of incomplete evacuation for ≥ 25% of defecations iv. Sensation of anorectal obstruction/blockage for ≥ 25% of defecations
9. Subjects who meet the modified Rome IV criteria based on history must also demonstrate the following during the 2 week Screening Phase diary assessment period:

   a. < 3 CSBMs each week b. ≤ 4 SBMs each week c. BSFS of 6 or 7 in < 25% of SBMs d. One out of the following three: i. BSFS of 1 or 2 in ≥ 25% of defecations ii. A straining value recorded on ≥ 25% of days when a BM was reported iii. ≥ 25% of BMs result in a sense of incomplete evacuation

Exclusion Criteria:

1. Subject has not maintained a stable diet for ≥ 30 days prior to the Screening Call or is unwilling to maintain a stable diet during the study.
2. Subject has had a surgical procedure requiring general anesthesia < 60 days before the Screening Call.
3. Subject has had a colonoscopy in the past 30 days or is scheduled for colonoscopy within the next 4 months and is unable/unwilling to postpone until the completion of study participation.
4. Subject has a history of cancer (other than basal cell carcinoma of the skin) unless the malignancy has been in a complete remission without maintenance therapy (eg, chemotherapy, radiation, surgery) for ≥ 5 years prior to the Screening Call.
5. Subject has any acute or chronic concomitant illness that could confound outcome assessments for this study, including, but not limited to:

   1. Known history of ulcerative colitis, Crohn's disease, colon cancer, current stomach ulcers, pancreatitis, diverticulitis.
   2. Known history of acute or chronic HBV, HCV, or HIV infection.
   3. Known or suspected alcoholism, drug addiction, or significant drug abuse within 1 year of the Screening Call.
6. Subject has any known medical condition, clinical signs and symptoms, vital signs, abnormal laboratory, or other testing, considered clinically significant by the Investigator, that could interfere with the subject's participation in and completion of the study including, but not limited to:

   1. Uncontrolled hypertension.
   2. Diabetes uncontrolled by diet (ie, requiring oral medication or insulin).
   3. Previous anaphylactic reaction to any medication.
   4. History of adrenal disease, diabetic nephropathy, or gastroparesis.
   5. Uncontrolled hypothyroidism.
   6. Untreated mental disorder
   7. Spinal cord injury
7. Subject has a history of severe drug allergy or hypersensitivity, or known hypersensitivity to any of the study product excipients.
8. Subject has had a cerebrovascular event (stroke) or myocardial infarction (MI) in the last 6 months.
9. Subject has plans to travel outside the USA during the study period.
10. Subject has a disease or condition other than CIC that has been associated with or can cause constipation.
11. Subject has a structural abnormality of the GI tract, or disease or condition that can affect GI motility, or defecation.
12. History or presence of pseudo obstruction, colon cancer, malignant polyps, colitis, ischemic colitis, abdominal adhesions, intestinal ischemia, esophageal atresia, laxative or enema abuse, or pelvic floor dysfunction.
13. Subject has a current COVID 19 infection, or a history or a prior COVID 19 infection with ongoing symptoms suggestive of "Long COVID".
14. Subject has active peptic ulcer disease not adequately treated or not stable with therapy.
15. Subject is taking a pharmacologic treatment for gastroesophageal reflux disease (GERD)/reflux that has not been stable for 15 days before the Screening Call.
16. Subject has a history of substantiated (documented by computed tomography (CT) scan or hospitalization) diverticulitis, or any ongoing chronic condition (eg, chronic pancreatitis, polycystic kidney disease, endometriosis, ovarian cysts, or other) that may be associated with chronic abdominal pain or discomfort and might confound the assessments in this study during the 2 years prior to the Screening Call.
17. Subject has had a fecal impaction that required hospitalization or emergency room treatment < 3 months before the Screening Call.
18. Subject has a history of an eating disorder in the last 5 years.
19. Subject has had surgery that meets any of the following criteria:

    1. Gastric bypass surgery or invasive procedure for the treatment of obesity or surgery to remove a segment of the GI tract at any time prior to the Screening Call
    2. Subjects who have had a gastric band unless the band has been completely removed > 60 days before the Screening Call
    3. Open surgery of the abdomen, pelvis, or retroperitoneal structures within 6 months prior to the Screening Call
20. Laparoscopic appendectomy or cholecystectomy or other instrumentation of the bowel < 60 days before the Screening Call.
21. Subject meets the Rome IV criteria for IBS C. This includes subjects who report abdominal pain or discomfort for ≥ 1 day/week in the last 3 months, with symptom onset ≥ 6 months prior to diagnosis, and whose abdominal pain or discomfort is associated with ≥ 2 of the following symptoms:

    1. Related to defecation
    2. Associated with a change in frequency of stool
    3. Associated with a change in form (consistency) of stool
22. Subject has had a barium enema within 7 days of the Screening Call.
23. Subject reports a clinically significant finding on colonoscopy.
24. Subject has taken a protocol prohibited drug within 15 days of the Screening Call or is not willing to abide by the protocol restrictions regarding use of prohibited drugs. (ie, medications that are known to either relieve or to potentially exacerbate constipation).
25. Subject has taken antibiotics or narcotics within 60 days of the Screening Call
26. Subject has previously taken the study product at any time.
27. Subject reports the use of bisacodyl or other medication for constipation on > 2 days in either of the 2 weeks in the Screening Phase assessment period.
28. Subject will be ineligible for randomization if, during the 2 week Screening Phase assessment, he or she has failed to complete at least 6 of the 7 required daily 'Daily Bowel Movement and Symptoms Questionnaire' questionnaires in each of the 2 weeks.
29. Subject uses bisacodyl or other medication for constipation within 72 hours before the first dose of study product (PP Day 1), to avoid confounding the data collected in the first week of study product administration, particularly the time to first BM.
30. Subject uses any narcotic during the course of the study.

Concomitant Treatment and Study Restrictions:

Prohibited concomitant treatments and study restrictions during the study and during the indicated periods include:

1. Any investigational drug product, device, or biologic within 3 months or five half lives (whichever is longer) prior to the Screening Call.
2. Any prescription or nonprescription medication for CIC.
3. Any prescription medication that has a significant risk of producing constipation. (eg, prokinetics, metformin, systemic glucocorticosteroids, non steroidal anti inflammatory drugs, ketoconazole, anticholinergics, or misoprostol) throughout any phase of the study.
4. Use of enemas, suppositories, or stimulant laxatives to have a BM more than 2 days in any week during the Screening, Product/Placebo and Product Phases.
5. Use of manual manipulation to have a BM.
6. Use of colon prep or high colonic throughout any phase of the study.

Permitted concomitant treatments and study restrictions during the study and during the indicated periods include:

1. Regular intake of acetylsalicylic acid (ie, aspirin) at doses up to 162 mg/day is permitted.
2. Rescue medication will not be provided; however, subjects may use bisacodyl (preferred) or other medication for constipation when at least 72 hours have passed since their previous BM or when their symptoms become intolerable. Use must be documented with all other concomitant medication use.

Other medication considered necessary for the subject's safety and well being may be allowed at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2022-06-12 (Actual)

PRIMARY OUTCOMES:
Tolerability as assessed using a PRO questionnaire, a 4 question Daily BM Questionnaire | 8 weeks
  A Complete Spontaneous Bowel Movement (CSBM) is a Bowel Movement (BM) that occurs in the absence of laxative use within 24 hours of the BM and the patient reports a feeling of complete evacuation. Tolerability is defined as no overall worsening of constipation measurement scores after 8 weeks of taking the product or the placebo compared to baseline scores. More complete spontaneous bowel movements is better, fewer is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Swann, MD, Principal Investigator — Microbiome Health Sciences
Locations (1):
- Remote Study - by phone and online, Manassas, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers